CLINICAL TRIAL: NCT04510766
Title: Molecular Characterization of Solid Tumors and Lymphomas to Optimize the Drug Development Process and Patients Enrollment in Early Phase Clinical Trials
Brief Title: Tumor Molecular Profiling in Early Phase Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Ente Ospedaliero Cantonale, Bellinzona (Other); Istituto Cantonale di Patologia (Other)
Responsible Party: Sponsor
Other Study IDs: IOSI-USNF-001
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tumor tissue and liquid biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A: Upon confirmation of the suitability for NGS analysis of the selected tumor sample, tumor DNA will be extracted and molecular profile will be performed using the pan-cancer NGS Ion TorrentTM OncomineTM Comprehensive Assay v3 according to manufacturer's instructions
- Part B: FFPE tumor archival tissue will be used to perform RNA-Seq with NGS HTG EdgeSeq Oncology Biomarker Panel Assay using the HTG machine following the manufacture's protocol. Blood samples for "liquid biopsy" will be collected at two time points: 1) Any time after enrollment in an early clinical trial and before starting the investigational agent
  (1 x 10 ml blood sample in EDTA tube as source of normal DNA for comparative analysis; 2 x 10 ml blood samples in cell-free DNA BCT Tubes for ctDNA collection; 2) At the time of radiological or clinical tumor progression (2 x 10 ml blood samples in cell-free DNA BCT Tubes for ctDNA collection). Blood samples will be collected and stored to create a biobank of "liquid biopsy" for future analysis.

SUMMARY:
Prospective, single centre, non-interventional exploratory research project that will be conducted on biological material and health-related personal data collected.

DETAILED DESCRIPTION:
Single center, two-parts pilot, prospective study to assess the role of molecular tumor profiling in supporting patient enrollment in early phase clinical trials.

Part A: patients with solid tumors or lymphomas (n=40) who are potential candidates for early phase clinical trials will be offered to have their more recent archival tumor tissue analyzed for the presence of somatic genomic alterations with the pan-cancer NGS Ion TorrentTM OncomineTM Comprehensive Assay v3 platform.

Part B: patients who have been enrolled in early phase clinical trials (estimated number: 16-18) will have their archival tumor tissue assessed with HTG EdgeSeq Oncology Biomarker Panel Assay for RNA-Seq to explore gene expression signatures and blood collected and stored to create a repository of samples (¨liquid biopsy¨) for future research with the aim to investigate the mutational profile of ctDNA at baseline and the acquisition of new mutations at the time of disease progression as a consequence of treatment exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age at least 18 years.
2. Patients with histological diagnosis of advanced solid tumor or lymphoma who are potential candidates for early phase clinical trials.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
4. Live expectancy of at least 6 months.
5. Availability of FFPE archival tumor tissue from previous surgery or diagnostic biopsy adequate for molecular analysis.
6. Ability to understand the patient information and study consent. Signed and dated written informed consent must be available before performing any study-related procedure.
7. Willing and able to comply with study procedures

Exclusion Criteria:

1. Presence of any clinical (e.g. concomitant disease, clinically significant symptoms, or non-clinical (psychological or social) conditions that would not make the patient eligible for enrolment in an early phase clinical trial.
2. Any other active malignancy (other than the one for which the subject is being assessed for trial option) that is progressing or requiring active treatment with the exception of basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological diagnosis of advanced solid tumor or lymphoma who are potential candidates for early phase clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accrual rate in early phase clinical trials | Two years
  Number of patients with available molecular profile enrolled per year

SECONDARY OUTCOMES:
Clinical Outcome | Two years
  Response rate among patients with available molecular tumor profiling that have been enrolled in an early phase clinical trial
Number of successful NGS-based DNA analysis performed on archival tissue | Two years
  Type and frequency of mutations identified on archival tissue
Number of NGS-based RNA-seq samples analyzed | Two years
  Analysis performed on archival tissue
Rate of stored samples | Two years
  Number of blood samples collected and stored for ctDNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Colombo, MD, Principal Investigator — Oncology Institute of Southern Switzerlan
Locations (1):
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland